CLINICAL TRIAL: NCT03042624
Title: Efficacy of Fermented Rice Flour for the Treatment of Atopic Dermatitis: Randomized, Double-blind Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Gian Vincenzo Zuccotti, Professor of Pediatrics, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FERCT16
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Dermatitis, Atopic; Child; Infant
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Parallel-arm, Randomized, Double-blind Controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each treatment is numbered consecutively without any reference to the underlying randomization scheme, which is known only to the statistician who generated the list and to the technician who prepared the packages. The packages and their contents are indistinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented rice (Experimental): 7 g of fermented rice flour powder obtained from Lactobacillus paracasei CBA L74 to be diluted in milk or water
  Interventions: Dietary Supplement: Fermented rice
- Maltodextrins (Placebo Comparator): 7 g of maltodextrins powder to be diluted in milk or water
  Interventions: Dietary Supplement: Maltodextrins

INTERVENTIONS:
Dietary Supplement: Fermented rice — 7 g of powder obtained from Lactobacillus paracasei CBA L74
  Arms: Fermented rice
Dietary Supplement: Maltodextrins — 7 g of maltodextrins powder
  Arms: Maltodextrins

SUMMARY:
This trial aims at evaluating the efficacy of a fermented rice flour for the treatment of atopic dermatitis (AD).

The fermented rice flour, obtained from Lactobacillus paracasei CBA L74 (Heinz Italia SpA, Latina, Italy), does not contain live bacteria. Lactobacillus paracasei CBA L74 belongs to the list of microorganisms with qualified presumption of safety compiled by the European Food Safety Authority (EFSA), is tested for the absence of antibiotic resistance genes in accordance with EFSA, and is genetically characterized by repetitive extragenic palindromic polymerase chain reaction.

Using a repeated-measure cohort design, the investigators have recently shown that the administration of a fermented-rice flour obtained from Lactobacillus paracasei CBA L74 was associated with a decrease of the score for atopic dermatitis (SCORAD) in children with AD.

The present randomized, double-blind, controlled trial is aimed at testing whether the fermented rice flour obtained from Lactobacillus paracasei CBA L74 is effective in reducing SCORAD in children with moderate to severe AD using placebo as comparator.

DETAILED DESCRIPTION:
Atopic dermatitis (AD), an itchy eczema with a chronic relapsing course, is the most common clinical manifestation of atopy in the first years of life.

On the basis of the available knowledge, AD is produced by an alteration of the skin barrier which triggers an inflammatory reaction. Such reaction is characterized by an early phase with abundance of Th2 cytokines (IL-4, IL-5) and eosinophils and by a later phase with predominance of Th1 cytokines (IL-2, IL-12 and IFN-gamma).

Emollients, possibly supplemented with ceramides, represent the first step of the treatment of AD. Corticosteroids are the most effective topical drugs. The use of topical immune-modulators (tacrolimus and pimecrolimus) offers an alternative to steroid therapy for long-term treatments. Severe cases require systemic therapy with steroids and cyclosporine and phototherapy with narrowband ultraviolet (UVB) and psoralen-ultraviolet A (PUVA) phototherapy.

The use of probiotics for the treatment of AD has attracted much interest in recent years but the available data are not conclusive. Probiotic-like effects can be obtained from inactivated bacteria or isolated bacterial components so that an extensive definition of probiotics has been proposed as bacterial cells or bacterial components that have a beneficial impact on the health and well-being of guests.

Using a repeated-measure cohort design, the investigators have recently shown that the administration of the fermented-rice flour obtained from Lactobacillus paracasei CBA L74 was associated with a decrease of SCORAD (score for atopic dermatitis) in children with AD.

SCORAD is the most commonly employed indicator of AD activity and its minimal clinically important difference is known, making it a suitable metric for clinical trials.

The fermented rice flour, obtained from Lactobacillus paracasei CBA L74 (Heinz Italia SpA, Latina, Italy), does not contain live bacteria. Lactobacillus paracasei CBA L74 belongs to the list of microorganisms with qualified presumption of safety compiled by the European Food Safety Authority (EFSA), is tested for the absence of antibiotic resistance genes in accordance with EFSA, and is genetically characterized by repetitive extragenic palindromic polymerase chain reaction.

Pre-clinical studies have shown anti-inflammatory effects of matrices fermented with Lactobacillus paracasei CBA-L74 in terms of production of IL-10 and reduction of IL-12 in response to bacterial stimulation. Such pre-clinical data were obtained on dendritic cells, on intestinal biopsies and on murine models.

The present randomized, double-blind, controlled trial is aimed at testing whether the fermented rice flour obtained from Lactobacillus paracasei CBA L74 is effective in reducing SCORAD in children with moderate to severe AD using placebo as comparator.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate or sever atopic dermatitis using SCORAD

Exclusion Criteria:

* acute rhino-conjunctivitis
* acute asthma
* autoimmune disease
* chronic obstructive pulmonary disease
* heart disease
* renal disease
* treatment with prebiotics 1 month before the enrolment
* treatment with probiotics 1 month before the enrolment
* treatment with antibiotics (undergoing)
* treatment with systemic immune-modulators 1 month before the enrolment
* treatment with local immune-modulators 1 month before the enrolment
* acute or chronic infectious disease
* known hypersensitivity to components of fermented rice flour

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-05-31 (Estimated)

PRIMARY OUTCOMES:
SCORAD change | 12 weeks
  The treatment will be stopped at 12 weeks

SECONDARY OUTCOMES:
SCORAD change | 16 weeks
  The outcome will be evaluated also 4 weeks after the suspension of treatment

OTHER OUTCOMES:
Fecal microbiota composition | 12 weeks
Cytokine profiling | 12 weeks
  Measurement of peripheral IFN-gamma, IL-4, IL-5, IL-10, IL-12, IL-13, IL-18 and IL-31
Peripheral immunophenotyping | 12 weeks
  Measurement of peripheral Treg, central memory and effector and Th1/Th2/Th17 cells
Total and specific IgE | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gian Vincenzo Zuccotti, MD, Principal Investigator — Pediatrics Department Ospedale dei Bambini V. Buzzi Milano
Locations (1):
- Pediatrics Department Ospedale dei Bambini V. Buzzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elias PM, Steinhoff M. "Outside-to-inside" (and now back to "outside") pathogenic mechanisms in atopic dermatitis. J Invest Dermatol. 2008 May;128(5):1067-70. doi: 10.1038/jid.2008.88. PMID 18408746
- [Background] Majamaa H, Isolauri E. Probiotics: a novel approach in the management of food allergy. J Allergy Clin Immunol. 1997 Feb;99(2):179-85. doi: 10.1016/s0091-6749(97)70093-9. PMID 9042042
- [Background] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Background] Weston S, Halbert A, Richmond P, Prescott SL. Effects of probiotics on atopic dermatitis: a randomised controlled trial. Arch Dis Child. 2005 Sep;90(9):892-7. doi: 10.1136/adc.2004.060673. Epub 2005 Apr 29. PMID 15863468
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Agostoni C, Goulet O, Kolacek S, Koletzko B, Moreno L, Puntis J, Rigo J, Shamir R, Szajewska H, Turck D; ESPGHAN Committee on Nutrition. Fermented infant formulae without live bacteria. J Pediatr Gastroenterol Nutr. 2007 Mar;44(3):392-7. doi: 10.1097/01.mpg.0000258887.93866.69. PMID 17325568
- [Background] Zagato E, Mileti E, Massimiliano L, Fasano F, Budelli A, Penna G, Rescigno M. Lactobacillus paracasei CBA L74 metabolic products and fermented milk for infant formula have anti-inflammatory activity on dendritic cells in vitro and protective effects against colitis and an enteric pathogen in vivo. PLoS One. 2014 Feb 10;9(2):e87615. doi: 10.1371/journal.pone.0087615. eCollection 2014. PMID 24520333
- [Background] Beretta S, Fabiano V, Petruzzi M, Budelli A, Zuccotti GV. Fermented rice flour in pediatric atopic dermatitis. Dermatitis. 2015 Mar-Apr;26(2):104-6. doi: 10.1097/DER.0000000000000103. No abstract available. PMID 25757084
- [Background] Schram ME, Spuls PI, Leeflang MM, Lindeboom R, Bos JD, Schmitt J. EASI, (objective) SCORAD and POEM for atopic eczema: responsiveness and minimal clinically important difference. Allergy. 2012 Jan;67(1):99-106. doi: 10.1111/j.1398-9995.2011.02719.x. Epub 2011 Sep 27. PMID 21951293